CLINICAL TRIAL: NCT02967757
Title: In-market Utilisation of Liraglutide Used for Weight Management in Europe: a Retrospective Medical Record Review Study.
Brief Title: In-market Utilisation of Liraglutide Used for Weight Management in Europe
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: NN8022-4241; U1111-1185-3661 (Other: WHO); EUPAS16225 (Registry Identifier: EU PAS Register)
Record Dates: First submitted 2016-11-16; First posted 2016-11-18 (Estimated); Last update posted 2023-01-20 (Actual); Status verified 2023-01

CONDITIONS: Metabolism and Nutrition Disorder; Obesity
MeSH Terms: conditions — Nutrition Disorders; Obesity | interventions — Liraglutide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- liraglutide 3.0 mg / liraglutide 1.2 mg/1.8 mg
  Interventions: Drug: liraglutide

INTERVENTIONS:
Drug: liraglutide — Patients will be treated according to routine clinical practice at the discretion of the treating physician. The study will gather data over the course of routine treatment for liraglutide 3.0 mg and liraglutide 1.2 mg/1.8 mg treated patients

SUMMARY:
This study is conducted in Europe. The aim of this study is to investigate usage of liraglutide for weight management in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Initiation of liraglutide 3.0 mg / liraglutide 1.2 mg/1.8 mg (initiation is defined as no prescription of the same brand within the previous 12 months)
* Informed consent obtained before any study-related activities. Study-related activities are any procedures that are carried out as part of the study, including activities to determine suitability of the study

Exclusion Criteria:

-Patients or physicians who previously participated in interventional studies for liraglutide 3.0 mg / liraglutide 1.2 mg/1.8 mg will not be eligible to participate in the study -For the full study, sites and patients included in the pilot will be excluded

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This is a descriptive study designed to examine in-market utilisation of liraglutide; thus there will be no hypothesis testing and a power calculation is not applicable. 100 patients will be enrolled for the pilot study (50 in each country, ) and additionally 300 patients will be enrolled for the full study (150 in each country)
Sampling Method: Non-Probability Sample
Enrollment: 316 (Actual)
Dates: Start 2016-12-22 (Actual); Primary Completion 2019-05-28 (Actual); Study Completion 2019-05-28 (Actual)

PRIMARY OUTCOMES:
Number of patients with BMI above or equal to 30 kg/m^2 | Less than 6 months before date of first prescription
Number of patients with BMI above or equal to 27kg/m^2 and below 30 kg/m^2 and 1 or more comorbidity | Less than 6 months before date of first prescription
  Dysglycaemia (Type 2 Diabetes Mellitus [T2DM] or prediabetes), hypertension, dyslipidaemia, obstructive sleep apnoea, and/or other weight-related comorbidities
Number of patients with above or equal to 27 kg/m^2 and below 30 kg/m^2 and no comorbidities | Less than 6 months before date of first prescription
  Dysglycaemia (Type 2 Diabetes Mellitus [T2DM] or prediabetes), hypertension, dyslipidaemia, obstructive sleep apnoea, and/or other weight-related comorbidities.
Number of patients with BMI below 27 kg/m^2 | Less than 6 months before date of first prescription
Number of patients with BMI not measured | Within 6 months before date of the first prescription

SECONDARY OUTCOMES:
Number of patients with liraglutide 1.2 or 1.8 mg prescriptions with dose information of 3.0 mg per day | From date of first prescription until 24 months
Number of patients with liraglutide 1.2 or 1.8 mg prescriptions and indication of weight management | From date of first prescription until 24 months
Number of patients with liraglutide 3.0 mg prescriptions who have reached a dose of 3.0 mg | By 12 weeks after first prescription date
  While adhering to the dose escalation according to label
Number of patients with liraglutide 3.0 mg prescriptions and other GLP-1 receptor agonists prescribed during continued treatment with liraglutide 3.0 mg | From date of first prescription until 24 months
  Number of patients
Number of patients with continued treatment with liraglutide 3.0 mg | From date of first prescription until 0-6 weeks; 7-12 weeks; 13-18 weeks; 19-24 months
  Number of patients

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR,1452), Study Director — Novo Nordisk A/S
Locations (18):
- Germany (9):
  - Novo Nordisk Investigational Site, Bad Nauheim
  - Novo Nordisk Investigational Site, Bünde
  - Novo Nordisk Investigational Site, Essen
  - Novo Nordisk Investigational Site, Hamburg
  - Novo Nordisk Investigational Site, Kaiserslautern
  - Novo Nordisk Investigational Site, Mainz
  - Novo Nordisk Investigational Site, München
  - Novo Nordisk Investigational Site, Münster
  - Novo Nordisk Investigational Site, Ulm
- Italy (9):
  - Novo Nordisk Investigational Site, Catania
  - Novo Nordisk Investigational Site, Chieti
  - Novo Nordisk Investigational Site, Cremona
  - Novo Nordisk Investigational Site, Novara
  - Novo Nordisk Investigational Site, Pisa
  - Novo Nordisk Investigational Site, Potenza
  - Novo Nordisk Investigational Site, Roma
  - Novo Nordisk Investigational Site, Rome
  - Novo Nordisk Investigational Site, Siena

REFERENCES:
- [Result] Sbraccia P, Aberle J, Olsen AH, Rathor N, Major-Pedersen A. Investigating the potential non-authorized use of two different formulations of liraglutide in Europe: A real-world drug utilization study. Diabetes Obes Metab. 2023 Apr;25(4):985-991. doi: 10.1111/dom.14945. Epub 2023 Jan 23. PMID 36514273